CLINICAL TRIAL: NCT06107088
Title: A Proof-of-concept Study to Evaluate the Effect and the Tolerability of a Novel Combination of Lactase Enzyme and Ligilactobacillus Salivarius DSM 34078 in Individuals With Lactose Intolerance
Brief Title: Effect of a Combination of Lactase and L. Salivarius DSM 34078 in Individuals With Lactose Intolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novozymes A/S (Industry)
Collaborators: Analyze & Realize (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NZ-2021-11; NOZ-DK/021121 (Other: analyze & realize)
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Lactose Intolerance
Keywords: lactase; Ligilactobacillus salivarius; lactose intolerance; hydrogen breath test
MeSH Terms: conditions — Lactose Intolerance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Test product1 (Experimental): 1 capsule 'lactase-bacterial strain combination' and 1 capsule placebo, once a day, one week
  Interventions: Dietary Supplement: Active 2; Dietary Supplement: Placebo
- Test product2 (Experimental): 1 capsule lactase and 1 capsule bacterial strain, once a day, one week
  Interventions: Dietary Supplement: Active 1; Dietary Supplement: Active 3
- Comparator (Active Comparator): 1 capsule lactase and 1 capsule placebo, once a day, one week
  Interventions: Dietary Supplement: Active 1; Dietary Supplement: Placebo
- Placebo (Placebo Comparator): 2 capsules placebo, once a day, one week
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Active 1 — lactase enzyme
  Arms: Comparator; Test product2
Dietary Supplement: Active 2 — lactase-bacterial strain combination
  Arms: Test product1
Dietary Supplement: Active 3 — bacterial strain alone
  Arms: Test product2
Dietary Supplement: Placebo — placebo
  Arms: Comparator; Placebo; Test product1

SUMMARY:
The goal of this clinical trial is to test whether a new combination of lactase and bacterial strain (L. Salivarius DSM 34078) can provide longer lasting beneficial effects on lactose digestion and gastrointestinal symptoms compared to lactase alone in people with lactose intolerance.

DETAILED DESCRIPTION:
Participants will attend 3 visits (V0, V1, V2). Visit 0 is a screening/baseline visit (5 to 10 days before Visit 1), where participants will be checked for inclusion and exclusion criteria, and undergo a lactose challenge (drink a cup of lactose containing water) followed by a hydrogen breath test (HBT) and Carbohydrate Perception Questionnaire (CPQ) measured at intervals over 3 hours. At Visit 1, eligible participants are randomized into one of the four study arms: Lactase and bacterial strain combination in a capsule; lactase and bacterial strain combination in separate capsules, lactase only, or placebo. Each Visit 1 and Visit 2 takes about 8 hours, where participants take the investigational product (IP) before the first lactose challenge (with first HBT and first CPQ for 3 hours), followed by a 2-hour break with standardized meal provided, and undergo a second lactose challenge (with second HBT and second CPQ for another 3 hours). Visit 2 is scheduled one week after Visit 1, where participants take the IP once daily at home for a week and fill in a diary between Visit 1 and 2. Stool samples are collected at Visit 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women from 18 to 65 years old
2. Self-reported:

   * previously diagnosed lactose intolerance or
   * presumed lactose intolerance, defined as GI complaints upon intake of lactose-containing food/beverage (such as abdominal pain, distension, bloating, flatulence, nausea, diarrhea), when no lactase or lactase-containing product has been used by the subject
3. Lactose maldigestion, confirmed by hydrogen breath test during lactose challenge at V0 (increase in H2 concentration of ≥ 20 parts per million (ppm) compared to value at t=0, during first 3 hours upon challenge)
4. Generally in good health as per investigator's judgement
5. Subject's ability and agreement to comply with study procedures, in particular:

   1. to adhere to conditions prior to test days
   2. keep the habitual dietary habits and physical activity (except with regard to conditions prior to test days); however, the consumption of lactose-containing products between V1 and V2 should be encouraged
   3. to complete study visits as required
   4. to avoid the use of other products which may influence the GI complaints during the study
   5. to avoid the use of lactase during the study
   6. to complete the subject diary and study questionnaires (including the questions that require the use of the Visual Analogue Scale (VAS))
6. Women of childbearing potential:

   1. commitment to use appropriate contraception methods
   2. negative pregnancy testing (beta human chorionic gonadotropin test in urine)
7. Readiness not to participate in another clinical study during this study

Participation is based upon written informed consent by the participant following written and oral information by the investigator regarding nature, purpose, consequences and possible risks of the clinical study.

Exclusion Criteria:

1. Self-reported known allergy or hypersensitivity to any components of the investigational products and/or chlorhexidine and/or standardised on-site meal
2. Self-reported congenital lactase deficiency (CLD)
3. Self-reported galactosemia
4. Self-reported history and/or presence of relevant GI disease or digestion/absorption disorder (e.g. inflammatory bowel disease, coeliac disease, gastroenteritis, severe constipation etc.) except for irritable bowel syndrome ((IBS); this condition is acceptable)
5. Self-reported inexplicable weight loss (>5%) within the last 3 months prior to study
6. Pulmonary disease that may interfere with the HBT
7. Hospital Anxiety and Depression Scale (HADS) anxiety or depression score of ≥11 at V0
8. Patient Health Questionnaire for Somatization (PHQ-15) score ≥15 at V0
9. Self-reported history and/or presence of other clinically significant condition/disorder, which per investigator's judgement could interfere with the results of the study or the safety of the subject, e.g.:

   1. uncontrolled thyroid gland disorder
   2. uncontrolled hypertension
   3. diabetes mellitus
   4. immunodeficiency
   5. scleroderma
   6. any other relevant serious organ or systemic diseases (e.g. cardiovascular, liver, renal, malignant, psychiatric disease etc.)
10. Significant GI surgery (except cholecystectomy, appendectomy) within the last 6 months prior to or planned during the study
11. Smoking
12. Colonoscopy or colon cleaning procedure within the last 4 weeks prior to and during the study
13. Regular medication and/or supplementation within the last 4 weeks prior to and during the study:

    1. antibiotics
    2. probiotics
    3. for management of LI complaints or any other that could influence gastrointestinal functions (e.g. laxatives (including fermentable dietary fibers), opioids, systemic corticosteroids, anticholinergics, anti-diarrheals, spasmolytics, prokinetics etc.) as per investigator judgement; intake of lactase prior to study is allowed
14. Clinically relevant deviation of safety laboratory parameter(s) at V0
15. Women of child-bearing potential: pregnancy or nursing
16. History of or current abuse of drugs, alcohol or medication
17. Participation in another study during the last 30 days prior to and during the study
18. Any other reason for exclusion as per investigator's judgment, e.g. insufficient compliance with study procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Difference in change in concentration of breath hydrogen between Test product1 and Comparator at the second lactose challenge of Visit 2, compared to baseline (Visit 0) | one week
  Change in the hydrogen concentration in the breath after lactose challenge is measured as incremental area under the curve (iAUC) for a period of 180 minutes
Difference in change in concentration of breath hydrogen between Test product2 and Comparator at the second lactose challenge of Visit 2, compared to baseline (Visit 0) | one week
  Change in the hydrogen concentration in the breath after lactose challenge is measured as incremental area under the curve (iAUC) for a period of 180 minutes

SECONDARY OUTCOMES:
Difference in change in concentration of breath hydrogen between Test product1 and Placebo at the second lactose challenge of Visit 2, compared to baseline (Visit 0) | one week
  Change in the hydrogen concentration in the breath after lactose challenge is measured as incremental area under the curve (iAUC) for a period of 180 minutes
Difference in change in concentration of breath hydrogen between Test product2 and Placebo at the second lactose challenge of Visit 2, compared to baseline (Visit 0) | one week
  Change in the hydrogen concentration in the breath after lactose challenge is measured as incremental area under the curve (iAUC) for a period of 180 minutes
Difference in change in concentration of breath hydrogen between Test product1 and Comparator at the second lactose challenge of Visit 1, compared to baseline (Visit 0) | Day 1
  Change in the hydrogen concentration in the breath after lactose challenge is measured as incremental area under the curve (iAUC) for a period of 180 minutes
Difference in change in concentration of breath hydrogen between Test product2 and Comparator at the second lactose challenge of Visit 1, compared to baseline (Visit 0) | Day 1
  Change in the hydrogen concentration in the breath after lactose challenge is measured as incremental area under the curve (iAUC) for a period of 180 minutes
Difference in change in concentration of breath hydrogen between Test product1 and Placebo at the second lactose challenge of Visit 1, compared to baseline (Visit 0) | Day 1
  Change in the hydrogen concentration in the breath after lactose challenge is measured as incremental area under the curve (iAUC) for a period of 180 minutes
Difference in change in concentration of breath hydrogen between Test product2 and Placebo at the second lactose challenge of Visit 1, compared to baseline (Visit 0) | Day 1
  Change in the hydrogen concentration in the breath after lactose challenge is measured as incremental area under the curve (iAUC) for a period of 180 minutes
Difference in change in concentration of breath hydrogen between Test product1 and Comparator at the first lactose challenge of Visit 2, compared to baseline (Visit 0) | one week
  Change in the hydrogen concentration in the breath after lactose challenge is measured as incremental area under the curve (iAUC) for a period of 180 minutes
Difference in change in concentration of breath hydrogen between Test product2 and Comparator at the first lactose challenge of Visit 2, compared to baseline (Visit 0) | one week
  Change in the hydrogen concentration in the breath after lactose challenge is measured as incremental area under the curve (iAUC) for a period of 180 minutes
Difference in change in concentration of breath hydrogen between Test product1 and Placebo at the first lactose challenge of Visit 2, compared to baseline (Visit 0) | one week
  Change in the hydrogen concentration in the breath after lactose challenge is measured as incremental area under the curve (iAUC) for a period of 180 minutes
Difference in change in concentration of breath hydrogen between Test product2 and Placebo at the first lactose challenge of Visit 2, compared to baseline (Visit 0) | one week
  Change in the hydrogen concentration in the breath after lactose challenge is measured as incremental area under the curve (iAUC) for a period of 180 minutes
Difference in change in concentration of breath hydrogen between Test product1 and Comparator at the first lactose challenge of Visit 1, compared to baseline (Visit 0) | Day 1
  Change in the hydrogen concentration in the breath after lactose challenge is measured as incremental area under the curve (iAUC) for a period of 180 minutes
Difference in change in concentration of breath hydrogen between Test product2 and Comparator at the first lactose challenge of Visit 1, compared to baseline (Visit 0) | Day 1
  Change in the hydrogen concentration in the breath after lactose challenge is measured as incremental area under the curve (iAUC) for a period of 180 minutes
Difference in change in concentration of breath hydrogen between Test product1 and Placebo at the first lactose challenge of Visit 1, compared to baseline (Visit 0) | Day 1
  Change in the hydrogen concentration in the breath after lactose challenge is measured as incremental area under the curve (iAUC) for a period of 180 minutes
Difference in change in concentration of breath hydrogen between Test product2 and Placebo at the first lactose challenge of Visit 1, compared to baseline (Visit 0) | Day 1
  Change in the hydrogen concentration in the breath after lactose challenge is measured as incremental area under the curve (iAUC) for a period of 180 minutes
Difference in change in global score of Carbohydrate Perception Questionnaire (CPQ) between Test product1 and Comparator at the second lactose challenge of Visit 2, compared to baseline (Visit 0) | one week
  Global score of CPQ is calculated as the sum of individual gastrointestinal symptom score of pain, bloating, flatulence, nausea and diarrhoea, each of which is defined as score of change from the time point 0 min to the time point with the maximal value during the period of 180 min after a lactose challenge
Difference in change in global score of Carbohydrate Perception Questionnaire (CPQ) between Test product2 and Comparator at the second lactose challenge of Visit 2, compared to baseline (Visit 0) | one week
  Global score of CPQ is calculated as the sum of individual gastrointestinal symptom score of pain, bloating, flatulence, nausea and diarrhoea, each of which is defined as score of change from the time point 0 min to the time point with the maximal value during the period of 180 min after a lactose challenge
Difference in change in global score of Carbohydrate Perception Questionnaire (CPQ) between Test product1 and Placebo at the second lactose challenge of Visit 2, compared to baseline (Visit 0) | one week
  Global score of CPQ is calculated as the sum of individual gastrointestinal symptom score of pain, bloating, flatulence, nausea and diarrhoea, each of which is defined as score of change from the time point 0 min to the time point with the maximal value during the period of 180 min after a lactose challenge
Difference in change in global score of Carbohydrate Perception Questionnaire (CPQ) between Test product2 and Placebo at the second lactose challenge of Visit 2, compared to baseline (Visit 0) | one week
  Global score of CPQ is calculated as the sum of individual gastrointestinal symptom score of pain, bloating, flatulence, nausea and diarrhoea, each of which is defined as score of change from the time point 0 min to the time point with the maximal value during the period of 180 min after a lactose challenge
Difference in change in global score of Carbohydrate Perception Questionnaire (CPQ) between Test product1 and Comparator at the second lactose challenge of Visit 1, compared to baseline (Visit 0) | Day 1
  Global score of CPQ is calculated as the sum of individual gastrointestinal symptom score of pain, bloating, flatulence, nausea and diarrhoea, each of which is defined as score of change from the time point 0 min to the time point with the maximal value during the period of 180 min after a lactose challenge
Difference in change in global score of Carbohydrate Perception Questionnaire (CPQ) between Test product2 and Comparator at the second lactose challenge of Visit 1, compared to baseline (Visit 0) | Day 1
  Global score of CPQ is calculated as the sum of individual gastrointestinal symptom score of pain, bloating, flatulence, nausea and diarrhoea, each of which is defined as score of change from the time point 0 min to the time point with the maximal value during the period of 180 min after a lactose challenge
Difference in change in global score of Carbohydrate Perception Questionnaire (CPQ) between Test product1 and Placebo at the second lactose challenge of Visit 1, compared to baseline (Visit 0) | Day 1
  Global score of CPQ is calculated as the sum of individual gastrointestinal symptom score of pain, bloating, flatulence, nausea and diarrhoea, each of which is defined as score of change from the time point 0 min to the time point with the maximal value during the period of 180 min after a lactose challenge
Difference in change in global score of Carbohydrate Perception Questionnaire (CPQ) between Test product2 and Placebo at the second lactose challenge of Visit 1, compared to baseline (Visit 0) | Day 1
  Global score of CPQ is calculated as the sum of individual gastrointestinal symptom score of pain, bloating, flatulence, nausea and diarrhoea, each of which is defined as score of change from the time point 0 min to the time point with the maximal value during the period of 180 min after a lactose challenge
Difference in change in global score of Carbohydrate Perception Questionnaire (CPQ) between Test product1 and Comparator at the first lactose challenge of Visit 2, compared to baseline (Visit 0) | one week
  Global score of CPQ is calculated as the sum of individual gastrointestinal symptom score of pain, bloating, flatulence, nausea and diarrhoea, each of which is defined as score of change from the time point 0 min to the time point with the maximal value during the period of 180 min after a lactose challenge
Difference in change in global score of Carbohydrate Perception Questionnaire (CPQ) between Test product2 and Comparator at the first lactose challenge of Visit 2, compared to baseline (Visit 0) | one week
  Global score of CPQ is calculated as the sum of individual gastrointestinal symptom score of pain, bloating, flatulence, nausea and diarrhoea, each of which is defined as score of change from the time point 0 min to the time point with the maximal value during the period of 180 min after a lactose challenge
Difference in change in global score of Carbohydrate Perception Questionnaire (CPQ) between Test product1 and Placebo at the first lactose challenge of Visit 2, compared to baseline (Visit 0) | one week
  Global score of CPQ is calculated as the sum of individual gastrointestinal symptom score of pain, bloating, flatulence, nausea and diarrhoea, each of which is defined as score of change from the time point 0 min to the time point with the maximal value during the period of 180 min after a lactose challenge
Difference in change in global score of Carbohydrate Perception Questionnaire (CPQ) between Test product2 and Placebo at the first lactose challenge of Visit 2, compared to baseline (Visit 0) | one week
  Global score of CPQ is calculated as the sum of individual gastrointestinal symptom score of pain, bloating, flatulence, nausea and diarrhoea, each of which is defined as score of change from the time point 0 min to the time point with the maximal value during the period of 180 min after a lactose challenge
Difference in change in global score of Carbohydrate Perception Questionnaire (CPQ) between Test product1 and Comparator at the first lactose challenge of Visit 1, compared to baseline (Visit 0) | Day 1
  Global score of CPQ is calculated as the sum of individual gastrointestinal symptom score of pain, bloating, flatulence, nausea and diarrhoea, each of which is defined as score of change from the time point 0 min to the time point with the maximal value during the period of 180 min after a lactose challenge
Difference in change in global score of Carbohydrate Perception Questionnaire (CPQ) between Test product2 and Comparator at the first lactose challenge of Visit 1, compared to baseline (Visit 0) | Day 1
  Global score of CPQ is calculated as the sum of individual gastrointestinal symptom score of pain, bloating, flatulence, nausea and diarrhoea, each of which is defined as score of change from the time point 0 min to the time point with the maximal value during the period of 180 min after a lactose challenge
Difference in change in global score of Carbohydrate Perception Questionnaire (CPQ) between Test product1 and Placebo at the first lactose challenge of Visit 1, compared to baseline (Visit 0) | Day 1
  Global score of CPQ is calculated as the sum of individual gastrointestinal symptom score of pain, bloating, flatulence, nausea and diarrhoea, each of which is defined as score of change from the time point 0 min to the time point with the maximal value during the period of 180 min after a lactose challenge
Difference in change in global score of Carbohydrate Perception Questionnaire (CPQ) between Test product2 and Placebo at the first lactose challenge of Visit 1, compared to baseline (Visit 0) | Day 1
  Global score of CPQ is calculated as the sum of individual gastrointestinal symptom score of pain, bloating, flatulence, nausea and diarrhoea, each of which is defined as score of change from the time point 0 min to the time point with the maximal value during the period of 180 min after a lactose challenge

CONTACTS AND LOCATIONS:
Overall Officials: Liana Vismane, MD, Principal Investigator — analyze & realize GmbH
Locations (1):
- Analyze & Realize Study Center, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No